CLINICAL TRIAL: NCT04659759
Title: COVID-19 in Pregnancy: Utilizing Immunology Through Epidemiology to Improve Perinatal/Neonatal Outcomes
Brief Title: COVID-19 Pregnancy Related Immunological, Clinical and Epidemiological Factors and Perinatal Outcomes
Acronym: COVID-PRICE
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Nemours (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20F.1043
Record Dates: First submitted 2020-12-07; First posted 2020-12-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Maternal serum/plasma
    * SARS-CoV-2 serology
    * Cytokine/chemokine panel
  * Cord blood serum/plasm
    * SARS-CoV-2 serology
    * Cytokine/chemokine panel
    * DNA methylation, miRNA/mRNA exression
  * Breastmilk o SARS-CoV-2 serology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID-19 Positive: Patients diagnosed with COVID-19 during pregnancy or while breastfeeding
  Interventions: Other: COVID-19 exposure
- COVID-19 vaccine: Patients who receive COVID-19 vaccine during pregnancy or while breastfeeding
  Interventions: Biological: COVID-19 vaccine
- Controls: Reproductive age women exposed to COVID-19 vaccine
- Pregnant Control: Pregnant women who delivered at TJUH, COVID negative

INTERVENTIONS:
Other: COVID-19 exposure — COVID-19 exposure during pregnancy
  Groups: COVID-19 Positive
Biological: COVID-19 vaccine — Receipt of any COVID-19 vaccine
  Groups: COVID-19 vaccine

SUMMARY:
This is a prospective cohort study of pregnant patients at an urban academic center diagnosed with perinatal COVID-19 infection, followed up to 6 weeks postpartum.

DETAILED DESCRIPTION:
This proposal aims to provide a multi-faceted approach to addressing perinatal COVID-19 infection by (1) improving our understanding of SARS-CoV-2 antibody specificity and durability over the course of pregnancy/postpartum in mother/baby dyad (2) understanding the downstream implications of maternal systemic inflammatory response with COVID-19 infection through study of fetal inflammatory response, placental pathology, and perinatal outcomes, and (3) to evaluate the interplay between socioeconomic characteristics, COVID-19, and early neonatal outcomes. (4) Evaluate antibody generation and durability in pregnant/breastfeeding women who receive any form of the COVID-19 vaccine

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 in pregnancy or within 6 months post partum
* Planned delivery at Thomas Jefferson University Hospital

Exclusion Criteria:

* Declines routine COVID testing on admission
* In active labor/pain/otherwise unable to provide consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients diagnosed with COVID-19 at any point during pregnancy or within 6 weeks post partum
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Maternal COVID-19 serology (IgG and IgM) | 6 weeks post partum
  IgG/IgM time profile through pregnancy up to 6 weeks post partum for those exposed to COVID-19
Maternal/neonatal IgG and IgM concordance | Delivery
  IgG/IgM at delivery in mother/neonate through maternal and cord blood sampling
Maternal COVID serology time/profile following vaccination | 6 months
  Baseline, 1m, 3m, 6m post second vaccine dose
Breastmilk Serology | 6months
  Breastmilk IgG and IgA time profile following COVID vaccine in breastfeeding women

SECONDARY OUTCOMES:
Breastmilk Serology | Delivery
  COVID-19 IgG and IgA in breast milk
Breastmilk Serology | 6 weeks post partum
  COVID-19 IgG and IgA in breastmilk
Cytokine | Delivery
  Compare maternal COVID (+) and COVID (-) cytokine panel
Neonatal cytokine | Delivery
  Compare cordblood cytokine panel between COVID(+) and COVID (-) at delivery
COVID disease vs vaccination immune response | 6 months
  Compare maternal IgG concentration time/profile in those with COVID disease vs COVID vaccine
COVID vaccine in pregnant vs nonpregnant | 6 months
  Compare maternal IgG concentration/time profile in pregnant vs non-pregnant women with vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States